CLINICAL TRIAL: NCT05918484
Title: Usefulness of Intermittently Scanned Continuous Glucose Monitoring in the Diagnosis of Maturity-onset Diabetes of the Young (MODY) Patients
Brief Title: Usefulness of Continuous Glucose Monitoring in MODY Diagnosis
Acronym: UCMODY
Status: Completed | Type: Observational
Sponsor: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Other Study IDs: C-621
Record Dates: First submitted 2023-06-07; First posted 2023-06-26 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes; MODY
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Type 1 diabetes patients: All type 1 diabetes patients using intermittently scanned continuous glucose monitoring (isCGM) in Castilla-La Mancha (Spain).
  Interventions: Device: Intermittenly scanned continuous glucose monitoring; Other: MODY genetic diagnostic test

INTERVENTIONS:
Device: Intermittenly scanned continuous glucose monitoring — Use of Intermittenly scanned continuous glucose monitoring (FreeStyle Libre) and meeting the glycometric data criteria:
  * Time in range 70-180 mg/L >70%
  * Glycemic management index <7%
  * Coefficient of variation <36%
Other: MODY genetic diagnostic test — Those patients fulfilling the glycometric data criteria and with clinical MODY suspicion:
  * diagnosis before 35 years of age
  * first-degree family history of diabetes.
  * negative pancreatic autoimmunity (Ac GAD, IA-2A and Ac ZnT8)
  * preserved pancreatic beta cell function defined as C-peptide > 0.2 ng/mL in the presence of plasma glycemia >140 mg/dL).
  Those patients who meet the previous criteria will proceed to the MODY genetic diagnostic test.

SUMMARY:
Observational study about usefulness of intermittently scanned continuous glucose monitoring (isCGM) in the diagnosis of maturity-onset of the young (MODY) patients.

DETAILED DESCRIPTION:
Cross-sectional retrospective analysis of all patients with type 1 diabetes (T1D) in Castilla-La Mancha (south-central Spanish region) using intermittently scanned continuous glucose monitoring (isCGM). This study aimed to asses the usefulness of isCGM in the diagnosis of MODY patients that were previously wrongly diagnosed as T1D patients.

The following glycometrics were taking into account as MODY predictors: time in range (70-180 mg/dL >70%, Glucose Management Index <7% y Coefficient of variation <36%. Patient´s clinical records of subjects meeting these glycometric criteria were reviewed for clinical suspicious of MODY (diagnosis before 35 years of age, first-degree family history of diabetes, negative pancreatic autoimmunity, preserved pancreatic beta cell function. Those patients meeting isCGM and clinical suspicious criteria were offered a diagnostic test for MODY.

The relationship between the qualitative outcome variable (MODY presence) and the quantitative variables will be performed using Student's t-test and ANOVA in situations of good fit with normality, and the Mann Whitney U and Kruskal Wallis when there is not a good fit with normality, and the Mann Whitney U and Kruskal Wallis when there is not.A P value < 0.05 was considered statistically significant.

The protocol was approved by the reference Castilla-La Mancha Public Health Institute Ethic Committee.

ELIGIBILITY:
Inclusion Criteria:

* Presence of T1D.
* Age equal or higher than 18 years old.
* In treatment with isCGM system.
* Active data in Libreview.
* isCGM use >70% of the possible time of use (isCGM data quality criteria).
* Time in range >70%, glucose management index <7% and coefficiente of variation <36% in the last 14 days glucometric recording.

Exclusion Criteria:

* Not receiving treatment with isCGM.
* Diagnosis of T1D in the last three years.
* Gestation in progress or programmed pregnancy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All T1D patients using isCGM in Castilla-La Mancha Public Health Service
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Positive predictive value | 14 days
  Positive predictive value of the combination of the glucometric variables TIR>70%, GMI <7% and CV <36% in the diagnosis of MODY. Units % (min 0, max 100)
Negative predictive value | 14 days
  Negative predictive value of the combination of the glucometric variables TIR>70%, GMI <7% and CV <36% in the diagnosis of MODY. Units % (min 0, max 100)
Sensitive | 14 days
  Sensitive of the combination of the glucometric variables TIR>70%, GMI <7% and CV <36% in the diagnosis of MODY. Units % (min 0, max 100)
Specificity | 14 days
  Specificity of the combination of the glucometric variables TIR>70%, GMI <7% and CV <36% in the diagnosis of MODY. Units % (min 0, max 100)

SECONDARY OUTCOMES:
Percetage of wrongly diagnosed type 1 diabetes patients | 14 days
  To assess the percentage of MODY patients with misdiagnosis of DM1. Units % (min 0, max 100)
Time in range of interstitial glucose in MODY patients | 14 days
  To assess the percetage of time in range (70-180 mg/dL, 3.9-10 mmol/L) of interstitial glucose in patients finally diagnosed as MODY. Units % (min 0, max 100)
Time above range of interstitial glucose in MODY patients. | 14 days
  To assess the percentage of time above range (>180 mg/dL, >10 mmol/L) of patients finally diagnosed as MODY. Units % (min 0, max 100)
Time beloww range of interstitial glucose in MODY patients. | 14 days
  To assess the percentage of time bellow range (<70 mg/dL, <3.9 mmol/L) of patients finally diagnosed as MODY. Units % (min 0, max 100)
Coefficient of variation of interstitial glucose in MODY patients. | 14 days
  To assess the coefficient of variations of patients finally diagnosed as MODY. Units % (min 0, max 100)
isCGM daily scan frequency in MODY patients | 14 days
  To analyze the use of iCGM in patients finally diagnosed as MODY through daily frequency of scanning (number daily scans, min 0-max 100).
Percentage of iCGM in MODY patients | 14 days
  To analyze the percentage of iCGM use in patients finally diagnosed as MODY (% time in use, units %, mix 0- max 100).

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Moreno-Fernandez, PhD, Principal Investigator — SESCAM
Locations (9):
- Spain (9):
  - Albacete University Hospital, Albacete, Albacete
  - La Mancha-Centro Hospital, Alcázar de San Juan, Ciudad Real
  - Santa Barbara Hospital, Puertollano, Ciudad Real
  - Valdepeñas General Hospital, Valdepeñas, Ciudad Real
  - Virgen de la Luz University Hospital, Cuenca, Cuenca
  - Guadalajara University Hospital, Guadalajara, Guadalajara
  - Maria Jose Picon, Málaga, Malaga
  - Virgen del Prado Hospital, Talavera de la Reina, Toledo
  - Toledo University Hospital, Toledo, Toledo

IPD SHARING:
Plan to Share IPD: Yes
Under other researchers request.
Time Frame: 1 monty after requested.
Access Criteria: Under other researchers request and after the approval of all researchers.

REFERENCES:
- [Background] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- [Background] Holt RIG, DeVries JH, Hess-Fischl A, Hirsch IB, Kirkman MS, Klupa T, Ludwig B, Norgaard K, Pettus J, Renard E, Skyler JS, Snoek FJ, Weinstock RS, Peters AL. The Management of Type 1 Diabetes in Adults. A Consensus Report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2021 Nov;44(11):2589-2625. doi: 10.2337/dci21-0043. Epub 2021 Sep 30. PMID 34593612
- [Background] Tosur M, Philipson LH. Precision diabetes: Lessons learned from maturity-onset diabetes of the young (MODY). J Diabetes Investig. 2022 Sep;13(9):1465-1471. doi: 10.1111/jdi.13860. Epub 2022 Jun 16. PMID 35638342
- [Background] Broome DT, Pantalone KM, Kashyap SR, Philipson LH. Approach to the Patient with MODY-Monogenic Diabetes. J Clin Endocrinol Metab. 2021 Jan 1;106(1):237-250. doi: 10.1210/clinem/dgaa710. PMID 33034350
- [Background] Shields BM, Shepherd M, Hudson M, McDonald TJ, Colclough K, Peters J, Knight B, Hyde C, Ellard S, Pearson ER, Hattersley AT; UNITED study team. Population-Based Assessment of a Biomarker-Based Screening Pathway to Aid Diagnosis of Monogenic Diabetes in Young-Onset Patients. Diabetes Care. 2017 Aug;40(8):1017-1025. doi: 10.2337/dc17-0224. PMID 28701371